CLINICAL TRIAL: NCT01066468
Title: A Non-randomized, Open-label Study to Characterize the Pharmacokinetics (PK) of Glivec/Gleevec® (Imatinib Mesylate) in Pediatric (Age Range 1 to Less Than 4 Years) Patients With Chronic Myeloid Leukemia (CML) or Philadelphia Chromosome Positive Acute Lymphoblastic Leukemia (Ph+ ALL) or Other Glivec/ Gleevec® Indicated Hematological Disorders (HES, CEL, MDS/ MPN)
Brief Title: Glivec/Gleevec Pediatric (Age 1 to Less Than 4) PK Study in CML, Ph+ ALL Patients and Other Glivec/Gleevec® Indicated Hematological Disorders.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: CSTI571A2110; 2010-018418-53 (EudraCT Number)
Record Dates: First submitted 2010-02-09; First posted 2010-02-10 (Estimated); Last update posted 2012-03-13 (Estimated); Status verified 2012-03

CONDITIONS: Chronic Myeloid Leukemia (CML); Philadelphia Chromosome Positive Acute Lymphoblastic Leukemia (Ph+ ALL); Other Glivec/Gleevec Indicated Hematological Disorders (HES, CEL, MDS/ MPN)
Keywords: Chronic myeloid leukemia; CML; Philadelphia chromosome positive; acute lymphoblastic leukemia; PhGlivec,; Gleevec,; hypereosinophilic syndrome,; HES,; chronic eosinophilic leukemia,; CEL,; myelodysplastic syndrome,; MDS,; myeloproliferative disease,; MPD+ ALL
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Hypereosinophilic Syndrome; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Pdgfra-Associated Chronic Eosinophilic Leukemia; Myelodysplastic Syndromes; Myeloproliferative Disorders | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gleevec/Glivec (Experimental)
  Interventions: Drug: Gleevec/Glivec

INTERVENTIONS:
Drug: Gleevec/Glivec
  Other Names: STI571

SUMMARY:
This study will assess the pharmacokinetics of imatinib in pediatric patients ages 1 to <4 years of age to help develop dosing regimens

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be 1 to less than 4 years of age at study entry
2. Written informed consent must be signed by the patient's parent or legal guardian.
3. Patients must have the diagnosis of CML or Ph+ ALL
4. Lansky score must be ≥ 50 (Table7-2)
5. Patient must have adequate end organ function as defined by

   * Total bilirubin < 1.5 x ULN
   * SGPT (ALT) and SGOT (AST) < 2.5 x UNL
   * Creatinine < 1.5 x ULN

Exclusion Criteria:

1. Patients who have received drugs a) known to be metabolized by CYP3A4 or 3A5, b) are CYP inhibitors and inducers, within 2 weeks prior to Visit 2 (except for imatinib)
2. Patients who previously received radiotherapy to ≥ 25% of the bone marrow, with the exception of patients who received total body radiation as part of a preparatory regimen for hematopoetic stem cell transplant (HSCT)
3. Patients receiving antibacterial and antipyretic medication to treat active infection
4. Patients with International normalized ratio (INR) or partial thromboplastin time (PTT) > 1.5 x ULN, with the exception of patients on treatment with oral anticoagulants
5. Patients whose parents or legal guardians, in the opinion of the Investigator, were unlikely to comply with the protocol or safety monitoring requirements

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 1 Year to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2010-10; Primary Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Measure: Pharmacokinetic data o (CL/F (clearance) o V/F (Volume of distribution) o Tmax o Physiologically based pharmacokinetic (PBPK) parameters (plasma protein binding and α-1 acid glycoprotein concentration) | 2 PK sample collection within 21 days

SECONDARY OUTCOMES:
safety and tolerability of imatinib during the study period | study period of 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Moscow, Russia